CLINICAL TRIAL: NCT02546817
Title: Eliquis (Apixaban) Regulatory Postmarketing Surveillance In Real World Practice (rPMS) For Venous Thromboembolism (VTE) Treatment And Prevention Of Recurrent VTE
Brief Title: Eliquis (VTE Treatment and Prevention of Recurrent VTE) rPMS
Status: Completed | Type: Observational
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Other Study IDs: CV185-440
Record Dates: First submitted 2015-09-07; First posted 2015-09-11 (Estimated); Last update posted 2017-10-31 (Actual); Status verified 2017-10

CONDITIONS: Venous Thromboembolism
Keywords: Treatment; Tx; Prevent
MeSH Terms: conditions — Venous Thromboembolism

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: No

SUMMARY:
To assess the real-world safety/effectiveness of Eliquis in Korean venous thromboembolism (VTE) patients and patient characteristics that are associated with bleeding among patients taking Eliquis. To identify factors that might be associated with the safety and effectiveness profile in Korean VTE patients.

ELIGIBILITY:
Inclusion Criteria:

* Adult (≥19 years of age) patients who are initiating treatment with Eliquis for the treatment of VTE or prevention of recurrent VTE for the first time in accordance with the Korean package insert will be enrolled in the study

Exclusion Criteria:

* Patients with prior treatment with Eliquis before enrollment in this study
* Patients receiving Eliquis treatment for an indication not approved indication in Korea
* Patients meeting any of the following criteria will not be included in the study:

  i) Hypersensitivity to the active substance or to any of the excipients

ii) Clinically significant active bleeding

iii) Hepatic disease associated with coagulopathy and clinically relevant bleeding risk

iv) Patients with increased bleeding risk due to such as following diseases:

1. Recent gastrointestinal ulceration history
2. Recent intracranial or intracerebral haemorrhage history
3. Intraspinal or intracerebral vascular abnormalities
4. Recent brain, spinal or ophthalmic surgery history
5. Recent brain or spinal injury
6. Known or suspected oesophageal varices
7. Arteriovenous malformations
8. Vascular aneurysms
9. Patients with malignant neoplasms at high risk of bleeding

   * Concomitant treatment with any other anticoagulant agent:

i) Unfractionated heparin (UFH)

ii) Low molecular weight heparins (enoxaparin, dalteparin, etc)

iii) Heparin derivatives (fondaparinux, etc)

iv) oral anticoagulants (warfarin, rivaroxaban, dabigatran, etc) except under the circumstances of switching therapy to or from apixaban or when UFH is given at doses necessary to maintain a patent central venous or arterial catheter

* Patients with rare hereditary problems of galactose intolerance, the Lapp lactose deficiency or glucose-galactose malabsorption

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult (≥19 years of age) patients who are initiating treatment with Eliquis for the treatment of VTE or prevention of recurrent VTE for the first time
Sampling Method: Non-Probability Sample
Enrollment: 29 (Actual)
Dates: Start 2015-11-30 (Actual); Primary Completion 2017-09-29 (Actual); Study Completion 2017-09-29 (Actual)

PRIMARY OUTCOMES:
Safety of Eliquis in Korean VTE patients based on incidence of adverse events (AEs), serious adverse events (SAEs) | Approximately 2 years
Patient characteristics that are associated with bleeding among patients taking Eliquis | Approximately 2 years
  Patient Characteristics: Age, sex, weight, height, baseline blood pressure, baseline serum creatinine, baseline creatinine clearance, and device insertion history

SECONDARY OUTCOMES:
Effectiveness of Eliquis in Korean VTE patients based on proportion of patients with no evidence of VTE and occurrence of VTE | Approximately 2 years
  For VTE treatment: The proportion of patients with recurrent VTE at 24 weeks will be calculated. The incidence proportion will be estimated
  For prevention of recurrent VTE: The proportion of patients with recurrent VTE at 24 weeks, 52 weeks, and 104 weeks, will be calculated. The incidence proportion will be estimated
Effectiveness of Eliquis in Korean VTE patients based on proportion of patients with no evidence of VTE and occurrence of VTE | Approximately 2 years
  For VTE treatment: The proportion of patients with recurrent VTE at 24 weeks will be calculated. The 95% confidence intervals will be estimated
  For prevention of recurrent VTE: The proportion of patients with recurrent VTE at 24 weeks, 52 weeks, and 104 weeks, will be calculated. The 95% confidence intervals will be estimated

CONTACTS AND LOCATIONS:
Overall Officials: Bristol Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (1):
- Local Institution, Seoul, South Korea

REFERENCES:
- See also: Investigator Inquiry Form — http://www.bms.com/clinical_trials/Pages/Investigator_inquiry_form.aspx